CLINICAL TRIAL: NCT01106300
Title: Assessment of Peripheral Muscle and Bone Mass in the Critically Ill and Its Response to External Muscle Stimulation
Brief Title: Musculoskeletal Ultrasound Study in Critical Care: Longitudinal Evaluation
Acronym: MUSCLE
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: King's College London (Other); Imperial College London (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 09/0167
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2014-04

CONDITIONS: Critical Illness; Septic Shock; Trauma; Organ Failure
MeSH Terms: conditions — Critical Illness; Shock, Septic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — quadricep muscle biopsy, blood and urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multi-organ failure: Sedated ventilated patients in multi-organ failure
- Single-organ failure: Sedated ventilated patients in single organ failure

SUMMARY:
Each year, 110,000 English/Welsh patients are admitted to Intensive Care Units (ICU). Many face prolonged disability as a result. Over two thirds have moderate-extreme limitation in their usual activity a year later, and one-third are severely affected, being unable to continue "most activities," or to live independently. Quite why known- but severe muscle wasting isn't may play an important role. We hope to find out, measuring the degree of wasting in patients, and seeking potential causes. We shall also address the mechanism of wasting, which may reflect an altered balance of activity in muscle growth pathways and those that break muscle down. We'll do this by collecting data, taking regular blood tests, scanning the leg muscles with an ultrasound machine, and analysing small muscle samples. In addition, we'll accurately and objectively measure how impaired these patients become, using specialist questionnaires, special monitoring equipment, simple walking tests and occasional special ('Cardio-Pulmonary') exercise tests. We'll try to see how badly activity is limited, and tease out whether muscle weakness plays a significant role in this. Finally, keeping muscles working (hard to do when unconscious/drowsy/bed-bound) may maintain muscle mass, so we'll see whether maintaining muscle activity using painless electrical stimulation will help.

ELIGIBILITY:
Inclusion Criteria:

* Ventilated patients aged > 18 years likely to survive and remain ventilated for 48 hours and on ICU for 7 days will be recruited.

Exclusion Criteria:

* Those who are pregnant,
* Have active malignancy,
* Have primary muscle/bilateral lower limb disorders or
* Are unlikely to survive 48 hrs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All admission to CRitical care who are ventilated, and are likely to remain so for 48hrs or more AND remain on ITU for 7 days
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2009-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cross sectional area of Rectus Femoris | 10 days
  Loss of 15% of Cross sectional area over 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Montgomery, MD, Study Chair — University College, London; Nicholas Hart, PhD, Study Chair — Guy's & St Thomas' NHS Foundation Trust, Kings College London; Zudin Puthucheary, MRCP, Principal Investigator — University College London, Whittington Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - Whittington Hospital NHS Trust, London, London
  - Kings College Hospital, London, London
  - Guy's & St Thomas' NHS Foundation Trust, London

REFERENCES:
- [Background] Rawal J, McPhail MJ, Ratnayake G, Chan P, Moxham J, Harridge SD, Hart N, Montgomery HE, Puthucheary ZA. A pilot study of change in fracture risk in patients with acute respiratory distress syndrome. Crit Care. 2015 Apr 14;19(1):165. doi: 10.1186/s13054-015-0892-y. PMID 25888496
- [Background] Puthucheary ZA, Phadke R, Rawal J, McPhail MJ, Sidhu PS, Rowlerson A, Moxham J, Harridge S, Hart N, Montgomery HE. Qualitative Ultrasound in Acute Critical Illness Muscle Wasting. Crit Care Med. 2015 Aug;43(8):1603-11. doi: 10.1097/CCM.0000000000001016. PMID 25882765
- [Result] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Result] Puthucheary ZA, McPhail MJ, Hart N. Acute muscle wasting among critically ill patients--reply. JAMA. 2014 Feb 12;311(6):622-3. doi: 10.1001/jama.2013.285426. No abstract available. PMID 24519306
- [Derived] Puthucheary ZA, Astin R, Mcphail MJW, Saeed S, Pasha Y, Bear DE, Constantin D, Velloso C, Manning S, Calvert L, Singer M, Batterham RL, Gomez-Romero M, Holmes E, Steiner MC, Atherton PJ, Greenhaff P, Edwards LM, Smith K, Harridge SD, Hart N, Montgomery HE. Metabolic phenotype of skeletal muscle in early critical illness. Thorax. 2018 Oct;73(10):926-935. doi: 10.1136/thoraxjnl-2017-211073. Epub 2018 Jul 6. PMID 29980655
- [Derived] McNelly AS, Rawal J, Shrikrishna D, Hopkinson NS, Moxham J, Harridge SD, Hart N, Montgomery HE, Puthucheary ZA. An Exploratory Study of Long-Term Outcome Measures in Critical Illness Survivors: Construct Validity of Physical Activity, Frailty, and Health-Related Quality of Life Measures. Crit Care Med. 2016 Jun;44(6):e362-9. doi: 10.1097/CCM.0000000000001645. PMID 26974547